CLINICAL TRIAL: NCT02992626
Title: Influence of Interacting With Dogs on Learning in Children
Brief Title: Influence of Dogs on Learning in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Tropical & Public Health Institute (Other)
Collaborators: University of Basel (Other)
Responsible Party: Principal Investigator, Karin Hediger, Principal Investigator, Swiss Tropical & Public Health Institute
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HAI1
Record Dates: First submitted 2016-12-12; First posted 2016-12-14 (Estimated); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Learning; Human-animal Interaction
MeSH Terms: conditions — Human-Animal Interaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- starting with dog (Experimental): Participants in this arm complete the first session in the presence of a dog. The second session is under control condition in the presence of a stuffed toy dog.
  Interventions: Other: Human-dog interaction; Other: Stuffed toy dog
- starting with control (Experimental): Participants in this arm complete the first session under control condition in the presence of a stuffed toy dog while the second session the tests are completed in the presence of a dog.
  Interventions: Other: Human-dog interaction; Other: Stuffed toy dog

INTERVENTIONS:
Other: Human-dog interaction — The tests are completed in the presence of a dog. Further, before starting the tests, the children have 15 minutes to interact with the present dog.
Other: Stuffed toy dog — The tests are completed in the presence of a stuffed toy dog. Further, before starting the tests, the children have 15 minutes to play with the stuffed toy dog.

SUMMARY:
In a randomised controlled cross-over study, the influence of interacting with a dog on children's learning performance is investigated.

ELIGIBILITY:
Inclusion Criteria:

* healthy
* 7 - 14 years old
* willingness to participate

Exclusion Criteria:

* medical or psychiatric diagnosis
* medication
* allergia (dogs)
* phobia (dogs)

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2016-05; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
VLMT (Verbaler Lern- und Merkfähigkeitstest) | 20 Minutes
  Number of remembered items within the test

SECONDARY OUTCOMES:
Digit Span (from HAWIK-IV) | 5 Minutes
  Number of remembered items (auditively presented numbers)
motoric task (from Kaufman Assessment Battery for Children, dt. Version (K-ABC)) | 5 Minutes
  Number of remembered items (visually presented gestures) that can be reproduced.
Heart rate/heart rate variability | 60 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hediger, Dr., Study Director — Swiss TPH / University of Basel
Locations (1):
- Aachen, Germany